CLINICAL TRIAL: NCT04681326
Title: PROPHYlactic Implantation of BIOlogic Mesh in Peritonitis: a Prospective Multicentric Randomized Controlled Trial
Brief Title: Prophylactic Implantation of Biologic Mesh in Peritonitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliero-Universitaria di Parma (Other)
Responsible Party: Principal Investigator, Fausto Catena, Director of Emergency and Trauma Surgery, Maggiore Hospital, Parma, Italy, Azienda Ospedaliero-Universitaria di Parma
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 506/2019/DISP/AOUPR
Record Dates: First submitted 2020-12-08; First posted 2020-12-23 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Incisional Hernia; Peritonitis
MeSH Terms: conditions — Incisional Hernia; Peritonitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biological prosthesis (Experimental): The subcutaneous tissue will be dissociated from the anterior rectum-muscles fascia to allow the positioning of the transfix stitches necessary to the mesh fixation. Successively the retro-muscular rectum muscles plane will be prepared by the separation of the rectum muscles from the posterior rectum-muscles fascia. The mesh will be fixed with at least 8 long-lasting absorbable transfix stitched placed at the cardinal and inter-cardinal points. The prosthesis will be placed with a 5 cm overlap. If the peritoneal plane can be sutured a Jackson-Pratt (JP) 10 suction drain will be placed under the prosthesis. A JP 10 suction drain will always be placed over the prosthesis. Anterior rectum fascia will be closed by emi-continuous monofilament suture with an intermediate- reabsorbable-time suture. Another JP 10 suction drain will be placed over the anterior fascia. No subcutaneous suture. Skin stapler or interrupted stitches will be used to close.
  Interventions: Device: biological prosthesis
- Standard of care (No Intervention): Normal abdominal wall closure

INTERVENTIONS:
Device: biological prosthesis — retro-muscular positioning of a swine dermal collagen prosthesis
  Arms: Biological prosthesis

SUMMARY:
Patients undergoing emergency surgery for peritonitis are at increased risk of abdominal wall-related complications. In patients with peritonitis the risk of incisional hernia (IH) is extremely elevated. The incidence of IH in patients operated with peritonitis is up to 54 %, compared with an incidence of 11-26 % in the general surgical population. Moreover, up to 24.1 % of patients with peritonitis undergoing emergency laparotomy may develop fascial dehiscence. The evaluation of quality of life of patients with IH showed lower mean scores on physical components of health-related quality of life and body image. The prophylactic mesh implantation demonstrated to reduce the incisional hernia rate in patients undergoing vascular or bariatric procedures. However, the intraperitoneal non absorbable mesh implantation in infected fields is generally considered at least of doubtful safety because of the theoretical increased risk of chronic mesh infection and enterocutaneous fistula. Most incisional hernias develop during the first three months after surgery, which represents the critical period for the healing of transected muscular and fibrous layers of the abdominal wall. However, most studies recommended a long-term follow up period of up to at least 5 years for midline abdominal incisions to determine the real incisional hernia rate. The midline abdominal incision is preferred in abdominal surgery, as it provides wide and rapid access compared other incisions. However, the incidence of incisional hernias is higher following midline abdominal incisions than in other abdominal incisions. In emergency surgery the midline incision in the majority of cases is a necessity. Several factors affect the process of wound healing: surgical site infection, poor surgical technique, and patient-related factors (i.e. peritonitis, old age, obesity, diabetes mellitus, nutritional deficiencies, hepatic cirrhosis, jaundice, renal impairment, malignancy, cardiac disease, chest problems, previous abdominal incisions, steroid therapy). Data about the use of biological prosthesis in infected fields are scarce and derive principally from case reports and case series. However, indications about their use and usefulness in infected fields have been recently published by the Italian Biological Prosthesis Working Group (IBPWG). A previously published prospective observational study evaluated the efficacy of implantation of biological prosthesis in high risk patients in order to reduce the incidence of incisional hernia. This study suggested the efficacy of this kind of prosthesis in reducing incisional hernia rate in patients with multiple risk factors. A recently published meta-analysis showed as the use of biological prosthesis in ventral hernia repair resulted in a lower infectious wound complication rate but in an similar recurrence rate. These results supports the application of biological prosthesis in high risk patients. One recent systematic review evaluated the positive effect on incisional hernia rate of the prophylactic mesh positioning in high risk patients. No randomized trials have been published since now about the use of biological prosthesis in contaminated or infected fields. The rationale of the trial is to evaluate the efficacy of the use of swine dermal collagen prosthesis implanted preperitoneally as a prophylactic procedure against incisional hernia in patients operated in urgency/emergency setting in contaminated/infected fields with peritonitis. The aim of the study is to reduce the incidence of incisional hernia from 50% to 20%.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged > 18 years old
* Clinical and/or laboratory and/or radiological evidence/signs of peritonitis of any origin (peritoneal reactivity, positive Blumberg sign, fever, free air/fluid in abdominal cavity, leucocytosis, increased C-Reactive Protein (CRP), lactic dehydrogenase (LDH), tachycardia, tachypnea, clinical or radiological evidence/suspect of bowel ischemia)
* Eventual strong suspect of possible bacterial translocation (reduction of the natural intestinal barrier against bacterial translocation, i.e. bowel ischemia, bowel overdistension, intestinal occlusion, etc.)
* Surgical indication for midline laparotomy independently from eventual previous laparotomies
* Informed consent

Exclusion Criteria:

* Patients aged < 18 years old
* Informed consent refusal
* No Clinical and/or laboratory and/or radiological evidence/signs of peritonitis of any origin
* Surgical indication for laparotomies other than midline one
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with incisional hernia | 3 months post surgery
  Comparison between number of patients with incisional hernia after surgery in the two arms of the study
Number of participants with incisional hernia | 6 months post surgery
  Comparison between number of patients with incisional hernia after surgery in the two arms of the study
Number of participants with incisional hernia | 12 months post surgery
  Comparison between number of patients with incisional hernia after surgery in the two arms of the study

SECONDARY OUTCOMES:
Incidence of adverse events after surgery for peritonitis | 3 months post surgery
  Number of patients with adverse events (prosthesis rejection, infection, seroma), after pre-peritoneal positioning of the swine dermal collagen prosthesis as prophylaxis for incisional hernia in peritonitis patients
Incidence of adverse events after surgery for peritonitis | 6 months post surgery
  Number of patients with adverse events (prosthesis rejection, infection, seroma), after pre-peritoneal positioning of the swine dermal collagen prosthesis as prophylaxis for incisional hernia in peritonitis patients
Incidence of adverse events after surgery for peritonitis | 12 months post surgery
  Number of patients with adverse events (prosthesis rejection, infection, seroma), after pre-peritoneal positioning of the swine dermal collagen prosthesis as prophylaxis for incisional hernia in peritonitis patients

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera-Universitaria di Parma, Parma, Italy

IPD SHARING:
Plan to Share IPD: No
The study result will be used for oral presentation, publications and seminars. The personal patient's data will be not share for privacy.

REFERENCES:
- [Derived] Coccolini F, Tarasconi A, Petracca GL, Perrone G, Giuffrida M, Disisto C, Sartelli M, Carcoforo P, Ansaloni L, Catena F. PROPHYlactic Implantation of BIOlogic Mesh in peritonitis (PROPHYBIOM): a prospective multicentric randomized controlled trial. Trials. 2022 Mar 4;23(1):198. doi: 10.1186/s13063-022-06103-4. PMID 35246206